CLINICAL TRIAL: NCT03690700
Title: The Feasibility and Effects of Low-load Blood-flow Restricted Exercise Following Spinal Cord Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Spinal Cord Injury Centre of Western Denmark (Other)
Collaborators: University of Southern Denmark (Other); Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Jørgen Feldbæk Nielsen, Research Director, Professor; PhD, Spinal Cord Injury Centre of Western Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BFRE_SCI
Record Dates: First submitted 2018-09-20; First posted 2018-10-01 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Spinal Cord Injuries
Keywords: BFR Exercise; Spinal Cord Injury; Neuromuscular Recovery; Randomized controlled study; Physical Function
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: randomized placebo controlled parallel group study
Who Masked: Participant
Masking Description: Prior to the first training session, participants will be block-randomized to either active BFRE (n=12) or sham BFRE (n=12), (control for gender). The participants will be blinded from the randomization
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- active BFRE (Active Comparator): 14 consecutive SCI patients are block-randomized to active arm
  Interventions: Other: BFRE
- sham BFRE (Sham Comparator): 14 consecutive SCI patients are block-randomized to sham arm
  Interventions: Other: BFRE

INTERVENTIONS:
Other: BFRE — BFR will be performed in the aBFRE group by use of pneumatic occlusion cuffs placed proximally on the thigh close to the inguinal fold, using an occlusion pressure corresponding to 40 % of seated arterial occlusion pressure (AOP). The individual AOP will be documented at baseline using doppler ultrasound (Siemens ACUSON S2000TM). Previous studies have shown that this pressure level can promote significant muscle adaptations to a similar degree and are associated with significantly less discomfort than higher occlusion pressures. The occlusion pressure of the participants in sham BFRE group will be 10mmHg.

SUMMARY:
Spinal cord injury (SCI): The World Health Organization estimates an incidence of 250,000 to 500,000 per year worldwide. In Denmark 130 new cases of SCI per year. SCI is a devastating condition: paresis/paralysis of the skeletal muscles below the injury site, partial or complete inability to walk, move and/or feel. Other sequelae are: infections, lifestyle diseases (cardiovascular, diabetes, nephrologic disease), mental wellbeing/suicide-risk profoundly raised , quality of life, next-of-kin affection. Recovery of motor function is high clinical priority and crucial for improved ADL outcomes. Strength training regimens have shown improved muscle strength in healthy subjects using near-maximal voluntary effort contractions, and few studies have demonstrated similar effects in a SCI population. Atrophy and fatigability and spasticity may reduce practical implementation for rehabilitation. Therefore, low-load blood-flow restricted exercise (BFRE) may prove beneficial as supplement to traditional rehabilitation, increasing muscle strength and inducing hypertrophy in healthy persons. BFRE is performed as low-intensity strength training (20-30 % of max) while simultaneously involving the use of circumferential placement of cuffs during exercise, to maintain arterial inflow to the muscle while preventing venous return. Based on existing scientific evidence, BFRE is acknowledged as a safe regime without serious side effects. Previously, the method has shown increased muscle strength and inducing skeletal muscle hypertrophy in addition to improvement in gait performance in individuals with various diseases causing reduced mobility. Purposes of this PhD project: to investigate the feasibility and effects of BFRE in individuals living with the consequences of SCI.

DETAILED DESCRIPTION:
BACKGROUND Spinal cord injury (SCI) represents a major health concern; the World Health Organization estimates an incidence of 250,000 to 500,000 per year worldwide. On average in Denmark we register 130 new cases of SCI per year. SCI is a devastating condition, in which paresis/paralysis of the skeletal muscles below the injury site results in a partial or complete inability to walk, move and/or feel. Concurrent to functional disabilities, infections, lifestyle diseases such as cardiovascular diseases are frequent sequelae due to inactivity and overweight. Affecting primarily younger and previously healthy individuals traumatic SCI also profoundly impacts the mental wellbeing of the patients and also their next-of-kin; quality of life (QoL) suffers and subsequently the risk of suicide for patients with SCI increases by two to five times as compared to the background population.

While a substantial effort is being put into the rehabilitation of individuals with SCI, large gaps in knowledge still exist on this area. Recovery of motor function is of high clinical priority as it is fundamental for improved ADL outcomes.

While various strength training regimens have been shown to increase muscle strength in neurologically intact individuals using near-maximal voluntary effort contractions, few studies have demonstrated similar effects from strength training regimens in persons with SCI. Complications such as atrophy and easily fatigable neuromuscular system with various degrees of spasticity often make these kinds of regimes less practical and rewarding for rehabilitation. Therefore, the addition of low-load blood-flow restricted exercise (BFRE) may prove beneficial as a supplement to traditional rehabilitation. Notable, BFRE is found to increase muscle strength and induces skeletal muscle hypertrophy in healthy individuals. Typically, BFRE is performed as low-load strength training (20-30 % 1 Repetition Maximum (RM)) combined with concurrent partial occlusion of limb blood flow by means of pneumatic cuffs placed proximal at the limb, to restrit arterial inflow to the exercising muscle and preventing venous return. Based on existing scientific evidence and applying pre-exercisescreening for known risk factors such as vascular dysfunction (AD) or prior history of trombosis, BFRE is acknowledged as a safe exercise regime without serious side effects. Previously, the method has shown increased muscle strength and skeletal muscle hypertrophy in addition to improvements in gait and sit-to-stand performance in individuals with various diseases causing reduced mobility.

The aim of this PhD project is to;

1. To conduct a pilot study for investigate the safety and feasibility of low-load BFRE training in adults with SCI
2. To conduct a RCT to investigate the effects of low-load blood-flow restricted exercise (BFRE) on physical function and neuromuscular recovery in individuals with SCI

The hypotheses are as following;

* The BFRE training protocol will be safe and applicable to individuals with a spinal cord injury
* Participants randomized to active BFRE treatment will exhibit greater increases in physical function and lower extremity muscle strength and muscle volume, respectively, than participants receiving sham BFRE. Treatment effects will be documented using functional disability assessment tools combined with measurements of maximum voluntary isometric muscle strength, rapid force capacity (rate of force development: RFD) and cross sectional area of the trained muscles.
* Participants allocated to active BFRE will exhibit less neuropathic pain than participants receiving sham BFRE. This will be documented by standardized questionnaires.

Feasibility Study (Study I)

The feasibility study will be conducted by the applicant, Anette Bach Jønsson (ABJ). Consecutively, prior to the RCT, 3 individuals with a SCI will be recruited between 1/4 2020 - 31/7 2021 using the same recruitment strategy and in- and exclusions criteria as in the RCT. Additionally, 3 in-patients with sub-acute SCI (Time since injury > 1 month and > 1 year) will be recruited. The 6 patients will follow the same initial examination and training protocol as in the active BFRE group as described below. However, the training will be performed twice a week for 2 weeks.

Outcome variables:

The following outcome measurements will be performed at pre- and postintervention.

Muscle testing Maximum, voluntary, isometric muscle strength that participants are able to exert on a portable knee dynamometer (S2P, Science to Practice, Ljubljana, Slovenia). Portable dynamometers are considered as valid and reliable instruments for measuring strength. Measurements of muscle torque (Nm) and Rate of Force Development (RFD, Nm/s) will be obtained.

Blood samples Blood samples will be obtained pre (30 minutes) and post (0-60 minutes) the first and last training session (4 blood samples in total). In-house physicians or laboratory technician will be responsible for retrieving the blood samples. Markers of coagulation (fibrinogen and D-dimer), fibrinolysis [tissue plasminogen activator (tPA)] and inflammation [high sensitivity C-reactive protein (hsCRP)] will be analyzed. The blood samples will be destroyed immediately after analyzing. The results will be obtained through the electronic patient record.

Feasibility Tolerance to the selected occlusion pressure and pain perception throughout training will be obtained by using the Numeric Rating Scale (NRS 0-11 point) and interview. Adherence to the planned training scheme will as well be recorded.

Safety considerations Autonomic dysreflexia (AD) may be a potentially life-threatening condition for people with a high injury level (Th6 and above, Tetraplegia) and may be provoked by cutaneous stimulation such as pain. Therefore, patients at risk of AD will be excluded and the ISCOS Autonomic Standards Assesment Form will be fulfilled before and after completion.

Eligibility for inclusion will be approved by specialist neurologist. Training sessions are coordinated with the physician-on-call. To ensure patient safety blood pressure and heart rate will be measured throughout training and will be closely monitored. In case of serious adverse events the MD on duty will be contacted immediately. During study I and II regular safety meetings in the research group will be scheduled. If serious adverse events occurs in study I, a reconsideration of the design of study II would be necessary (e.g. changes in BFR-dosage) and further pilot testing would be necessary.

Randomized controlled trial (Study II)

Methods:

Initial examination:

After inclusion, medical history, demographic and anthropometric data, and the neurological level of SCI will be obtained. Information about the trauma and neurological level (masured by the International Standards for Neurological Classification of SCI (ISNCSCI)) will be obtained through the electronic patient record. Furthermore, functional disability assessment in addition to para-clinical tests will be conducted

Intervention/Control Prior to the first training session, participants will be randomized to either active BFRE (n=14) or sham BFRE (n=14), while controlling for gender. BFR will be performed in the aBFRE group by use of pneumatic occlusion cuffs placed proximally on the thigh close to the inguinal fold, using an occlusion pressure corresponding to 40 % of seated arterial occlusion pressure (AOP). The individual AOP will be documented at baseline using doppler ultrasound (Siemens ACUSON S2000TM). Previous studies have shown that this pressure level can promote significant muscle adaptations to a similar degree and are associated with significantly less discomfort than higher occlusion pressures. The occlusion pressure of the participants in sham BFRE group will be approx.10mmHg.

Subjects from both groups will participate in 45 minutes of low-intensity BFRE (30-40% 1RM) of the lower extremities twice/week for 8 weeks, consisting of 5 minutes light warm-up of low-intensity cycling followed by 4 sets (30x15x15x15 repetitions, 45 sec pause between sets) of seated leg extension and leg curl with BFR. A 3 minutes pause is allowed between exercises where the cuff will be deflated. Blood pressure will be measured before and after each completed exercise (5 measures in total per session).

Data analysis Within-group changes from baseline to follow-up will be analyzed using paired parametric or nonpar-ametric methods. Between-group differences will be compared as unpaired data using a parametric or nonparametric methods. The type 1 level of significance is set at 0.05. The results will be analyzed according to the intention-to-treat principle. According to sample-size calculation with an 80 % power and 5 % level of significance a difference of 20 % on MVC between the active and sham BFR groups are possible to detect with 24 participants. A total of 28 participants will be recruited to take a 20 % dropout rate into account. A difference of 20 % on MVC is expected as a realistic suggestion as a minimal clinical important difference.

Practical framework This PhD project has received permission from SCIWDK. The initial examination and tests at baseline and follow-up will be conducted at SCIWDK's laboratory by the applicant, Anette Bach Jønsson (ABJ). She is an experienced physiotherapist. Training sessions will be guided and supervised by in-house physiotherapists and ABJ.

Ethical considerations:

The study has been approved by The Danish Scientific Ethics Commission (Ref No. 1-10-72-290-18), and by Data Protection Agency (Datatilsynet, Ref No. 1-16-02-640-18) and has been reported to Clinicaltrials.gov.

Economy: Not described here

ELIGIBILITY:
Inclusion Criteria:

* Duration of SCI > 1 year,
* 18 years of age or older
* Exhibit a grade 2, 3 or 4 muscle function of the knee flexors and/or extensors
* Classification of grades A, B, C or D on the International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) scale
* Cognitive ability to follow instructions

Exclusion Criteria:

* Substance abuse
* Severe mental illness
* Uncontrolled hypertension
* Severe arteriosclerosis, coronary arterial disease
* History of severe autonomic dysreflexia
* Deep venous thrombosis (or severe coagulation dysfunction)
* Collagen diseases such as Ehlers-Danlos Syndrome and Marfan's Syndrome
* Severe neuropathies

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Changes in MVC | 1 week before treatment; 4-, 8- and 12-weeks after start of treatment
  Changes in maximum, voluntary, isometric muscle strength (Muscle torque, MVC) of the m. quadriceps and hamstrings from baseline to follow-up

SECONDARY OUTCOMES:
Change in Rate of force development (RFD) | 1 week before treatment; 4-,8- and 12-weeks after start of treatment
  Rate of force development (RFD) measurements of the m. quadriceps and hamstrings
Change in muscle and tendon thickness | 1 week before treatment; 4-, 8- and 12-weeks after start of treatment
  Muscle and tendon thickness of the muscles in the upper leg
Change in The Spinal Cord Ability Ruler (SCAR) | 1 week before treatment; 4-, 8- and 12-weeks after start of treatment
  SCAR measures the performance of volitional tasks along with assessment of functional muscle contractions
Timed Up & Go Test (TUG) | 1 week before treatment; 4-, 8- and 12-weeks after start of treatment
  TUG is a standardized and reliable test for assessment of mobility, balance and walking ability in patients with SCI
Timed 10 Meter Walk Test | 1 week before treatment; 4-, 8- and 12-weeks after start of treatment
  Timed 10 Meter Walk Test assesses short duration walking speed. The tests has demonstrated an excellent reliability in patients with SCI
6 Minute Walk Test | 1 week before treatment; 4-, 8- and 12-weeks after start of treatment
  6 Minute Walk Test is a reliable and valid sub-maximal test of aerobic capacity/endurance
Walking Index for Spinal Cord Injury (WISCI-II) | 1 week before treatment; 4-, 8- and 12-weeks after start of treatment
  WISCI-II is a valid and reliable test, which assesses the type and amount of assistance required by a person with spinal cord injury (SCI) for walking
Change in self-reported, neuropathic pain level | 1 week before treatment; 4-, 8- and 12-weeks after start of treatment
  Numeric Rating Scale (NRS, scale 0-10) is a validated, subjective measure for acute and chronic neuropathic pain.
Changes in blood marker - Growth hormone, Insulin-like growth factor 1 (IGF-1), creatine kinase, cortisol, testosterone, myoglobin | Immediately before and three hours after the first training session. Additionally, 4-, 8- and 12-weeks after start of treatment
  Venous blood samples regarding muscle damage, recovery and protein synthesis will be obtained
Changes in quality of life | 1 week before treatment; 4-, 8- and 12-weeks after start of treatment
  International spinal cord injury data sets - quality of life basic data set (QoLBDS) is a short valid questionnaire investigating QoL in a SCI population
Changes in WHODAS 2.0 | 1 week before treatment; 4-, 8- and 12-weeks after start of treatment
  WHODAS 2.0 is a reliable and valid instrument measuring activity and participation in the context of functioning in people with SCI
Changes in accelerometer data | Accelerometer data will be obtained 3 x 1 week prior to and during the intervention period.
  Activity classification using accelerometers will be obtained using a sensor on the upper leg

CONTACTS AND LOCATIONS:
Overall Officials: Jørgen Feldbæk Nielsen, MD,PhD,Prof., Principal Investigator — Spinal Cord Injury Centre of Western Denmark
Locations (1):
- The Spinal Cord Injury Centre of Western Denmark, Viborg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reed R, Mehra M, Kirshblum S, Maier D, Lammertse D, Blight A, Rupp R, Jones L, Abel R, Weidner N; EMSCI Study Group; SCOPE; Curt A, Steeves J. Spinal cord ability ruler: an interval scale to measure volitional performance after spinal cord injury. Spinal Cord. 2017 Aug;55(8):730-738. doi: 10.1038/sc.2017.1. Epub 2017 Mar 21. PMID 28322239
- [Background] Aagaard P, Simonsen EB, Andersen JL, Magnusson P, Dyhre-Poulsen P. Increased rate of force development and neural drive of human skeletal muscle following resistance training. J Appl Physiol (1985). 2002 Oct;93(4):1318-26. doi: 10.1152/japplphysiol.00283.2002. PMID 12235031
- [Background] Gregory CM, Bowden MG, Jayaraman A, Shah P, Behrman A, Kautz SA, Vandenborne K. Resistance training and locomotor recovery after incomplete spinal cord injury: a case series. Spinal Cord. 2007 Jul;45(7):522-30. doi: 10.1038/sj.sc.3102002. Epub 2007 Jan 16. PMID 17228358
- [Background] Harvey LA, Fornusek C, Bowden JL, Pontifex N, Glinsky J, Middleton JW, Gandevia SC, Davis GM. Electrical stimulation plus progressive resistance training for leg strength in spinal cord injury: a randomized controlled trial. Spinal Cord. 2010 Jul;48(7):570-5. doi: 10.1038/sc.2009.191. Epub 2010 Jan 12. PMID 20065991
- [Background] Gorgey AS, Timmons MK, Dolbow DR, Bengel J, Fugate-Laus KC, Michener LA, Gater DR. Electrical stimulation and blood flow restriction increase wrist extensor cross-sectional area and flow meditated dilatation following spinal cord injury. Eur J Appl Physiol. 2016 Jun;116(6):1231-44. doi: 10.1007/s00421-016-3385-z. Epub 2016 May 7. PMID 27155846
- [Background] Pelletier CA, Hicks AL. Muscle fatigue characteristics in paralyzed muscle after spinal cord injury. Spinal Cord. 2011 Jan;49(1):125-30. doi: 10.1038/sc.2010.62. Epub 2010 Jun 8. PMID 20531355
- [Background] Slysz J, Stultz J, Burr JF. The efficacy of blood flow restricted exercise: A systematic review & meta-analysis. J Sci Med Sport. 2016 Aug;19(8):669-75. doi: 10.1016/j.jsams.2015.09.005. Epub 2015 Sep 28. PMID 26463594
- [Background] Loenneke JP, Wilson JM, Marin PJ, Zourdos MC, Bemben MG. Low intensity blood flow restriction training: a meta-analysis. Eur J Appl Physiol. 2012 May;112(5):1849-59. doi: 10.1007/s00421-011-2167-x. Epub 2011 Sep 16. PMID 21922259
- [Background] Takarada Y, Takazawa H, Sato Y, Takebayashi S, Tanaka Y, Ishii N. Effects of resistance exercise combined with moderate vascular occlusion on muscular function in humans. J Appl Physiol (1985). 2000 Jun;88(6):2097-106. doi: 10.1152/jappl.2000.88.6.2097. PMID 10846023
- [Background] Loenneke JP, Wilson JM, Wilson GJ, Pujol TJ, Bemben MG. Potential safety issues with blood flow restriction training. Scand J Med Sci Sports. 2011 Aug;21(4):510-8. doi: 10.1111/j.1600-0838.2010.01290.x. Epub 2011 Mar 16. PMID 21410544
- [Background] Cook SB, LaRoche DP, Villa MR, Barile H, Manini TM. Blood flow restricted resistance training in older adults at risk of mobility limitations. Exp Gerontol. 2017 Dec 1;99:138-145. doi: 10.1016/j.exger.2017.10.004. Epub 2017 Oct 5. PMID 28987643
- [Background] Ferraz RB, Gualano B, Rodrigues R, Kurimori CO, Fuller R, Lima FR, DE Sa-Pinto AL, Roschel H. Benefits of Resistance Training with Blood Flow Restriction in Knee Osteoarthritis. Med Sci Sports Exerc. 2018 May;50(5):897-905. doi: 10.1249/MSS.0000000000001530. PMID 29266093
- [Background] Jorgensen AN, Aagaard P, Nielsen JL, Frandsen U, Diederichsen LP. Effects of blood-flow-restricted resistance training on muscle function in a 74-year-old male with sporadic inclusion body myositis: a case report. Clin Physiol Funct Imaging. 2016 Nov;36(6):504-509. doi: 10.1111/cpf.12259. Epub 2015 Jun 19. PMID 26095885
- [Background] Itzkovich M, Gelernter I, Biering-Sorensen F, Weeks C, Laramee MT, Craven BC, Tonack M, Hitzig SL, Glaser E, Zeilig G, Aito S, Scivoletto G, Mecci M, Chadwick RJ, El Masry WS, Osman A, Glass CA, Silva P, Soni BM, Gardner BP, Savic G, Bergstrom EM, Bluvshtein V, Ronen J, Catz A. The Spinal Cord Independence Measure (SCIM) version III: reliability and validity in a multi-center international study. Disabil Rehabil. 2007 Dec 30;29(24):1926-33. doi: 10.1080/09638280601046302. Epub 2007 Mar 5. PMID 17852230
- [Background] Kirshblum SC, Waring W, Biering-Sorensen F, Burns SP, Johansen M, Schmidt-Read M, Donovan W, Graves D, Jha A, Jones L, Mulcahey MJ, Krassioukov A. Reference for the 2011 revision of the International Standards for Neurological Classification of Spinal Cord Injury. J Spinal Cord Med. 2011 Nov;34(6):547-54. doi: 10.1179/107902611X13186000420242. PMID 22330109
- [Background] Kalsi-Ryan S, Beaton D, Curt A, Duff S, Popovic MR, Rudhe C, Fehlings MG, Verrier MC. The Graded Redefined Assessment of Strength Sensibility and Prehension: reliability and validity. J Neurotrauma. 2012 Mar 20;29(5):905-14. doi: 10.1089/neu.2010.1504. Epub 2011 Aug 12. PMID 21568688
- [Background] Whitehurst DG, Engel L, Bryan S. Short Form health surveys and related variants in spinal cord injury research: a systematic review. J Spinal Cord Med. 2014 Mar;37(2):128-38. doi: 10.1179/2045772313Y.0000000159. Epub 2014 Jan 6. PMID 24559417
- [Background] Wressle E, Marcusson J, Henriksson C. Clinical utility of the Canadian Occupational Performance Measure--Swedish version. Can J Occup Ther. 2002 Feb;69(1):40-8. doi: 10.1177/000841740206900104. PMID 11852689
- [Background] Stark T, Walker B, Phillips JK, Fejer R, Beck R. Hand-held dynamometry correlation with the gold standard isokinetic dynamometry: a systematic review. PM R. 2011 May;3(5):472-9. doi: 10.1016/j.pmrj.2010.10.025. PMID 21570036
- [Background] Gorgey AS, Timmons MK, Michener LA, Ericksen JJ, Gater DR. Intra-rater reliability of ultrasound imaging of wrist extensor muscles in patients with tetraplegia. PM R. 2014 Feb;6(2):127-33. doi: 10.1016/j.pmrj.2013.08.607. Epub 2013 Sep 13. PMID 24041587
- [Background] Phadke CP, Robertson CT, Condliffe EG, Patten C. Upper-extremity H-reflex measurement post-stroke: reliability and inter-limb differences. Clin Neurophysiol. 2012 Aug;123(8):1606-15. doi: 10.1016/j.clinph.2011.12.012. Epub 2012 Jan 23. PMID 22277759
- [Background] Ansari NN, Naghdi S, Arab TK, Jalaie S. The interrater and intrarater reliability of the Modified Ashworth Scale in the assessment of muscle spasticity: limb and muscle group effect. NeuroRehabilitation. 2008;23(3):231-7. PMID 18560139
- [Background] Klomjai W, Katz R, Lackmy-Vallee A. Basic principles of transcranial magnetic stimulation (TMS) and repetitive TMS (rTMS). Ann Phys Rehabil Med. 2015 Sep;58(4):208-213. doi: 10.1016/j.rehab.2015.05.005. Epub 2015 Aug 28. PMID 26319963
- [Background] Maxwell L, Santesso N, Tugwell PS, Wells GA, Judd M, Buchbinder R. Method guidelines for Cochrane Musculoskeletal Group systematic reviews. J Rheumatol. 2006 Nov;33(11):2304-11. PMID 17086611
- [Background] Stavres J, Singer TJ, Brochetti A, Kilbane MJ, Brose SW, McDaniel J. The Feasibility of Blood Flow Restriction Exercise in Patients With Incomplete Spinal Cord Injury. PM R. 2018 Dec;10(12):1368-1379. doi: 10.1016/j.pmrj.2018.05.013. Epub 2018 May 23. PMID 29802910
- [Derived] Jonsson AB, Krogh S, Lillelund S, Aagaard P, Kasch H, Nielsen JF. Efficacy of Blood Flow Restriction Exercise for Improving Lower Limb Muscle Strength and Function in Chronic Spinal Cord Injury: A Randomized Controlled Trial. Scand J Med Sci Sports. 2024 Dec;34(12):e14759. doi: 10.1111/sms.14759. PMID 39636092
- [Derived] Jonsson AB, Krogh S, Severinsen KE, Aagaard P, Kasch H, Nielsen JF. Feasibility and safety of two weeks of blood flow restriction exercise in individuals with spinal cord injury. J Spinal Cord Med. 2026 Jan;49(1):58-67. doi: 10.1080/10790268.2024.2408052. Epub 2024 Oct 11. PMID 39392467